CLINICAL TRIAL: NCT00543387
Title: A Phase I Investigation of MK-5108 and MK-5108 With Docetaxel in Patients With Advanced Solid Tumors
Brief Title: Treatment of Participants With Advanced and/or Refractory Solid Tumors (MK-5108-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5108-001; 2007_598 (Other: Sponsor Registry Number); MK-5108-001 (Other: Merck Protocol Number)
Record Dates: First submitted 2007-10-12; First posted 2007-10-15 (Estimated); Results first posted 2018-11-09 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Cancer, Neoplasms, Tumors
MeSH Terms: conditions — Neoplasms | interventions — 4-(3-chloro-2-fluorophenoxy)-1-((6-(1,3-thiazol-2-ylamino)pyridin to 2-yl)methyl) cyclohexanecarboxylic acid; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (11):
- MK-5108 200 mg BID (Panel 1) (Experimental): Participants receive 200 mg of MK-5108 orally twice daily (BID) the first 2 days of a 14-day cycle (cycle extended to 21 days if ≥Grade 2 toxicity observed).
  Interventions: Drug: MK-5108
- MK-5108 400 mg BID (Panel 1) (Experimental): Participants receive 400 mg of MK-5108 orally BID the first 2 days of a 14-day cycle (cycle extended to 21 days if ≥Grade 2 toxicity observed).
  Interventions: Drug: MK-5108
- MK-5108 800 mg BID (Panel 1) (Experimental): Participants receive 800 mg of MK-5108 orally BID the first 2 days of a 14-day cycle (cycle extended to 21 days if ≥Grade 2 toxicity observed).
  Interventions: Drug: MK-5108
- MK-5108 1200 mg BID (Panel 1) (Experimental): Participants receive 1200 mg of MK-5108 orally BID the first 2 days of a 14-day cycle (cycle extended to 21 days if ≥Grade 2 toxicity observed).
  Interventions: Drug: MK-5108
- MK-5108 1500 mg BID (Panel 1) (Experimental): Participants receive 1500 mg of MK-5108 orally BID the first 2 days of a 14-day cycle (cycle extended to 21 days if ≥Grade 2 toxicity observed).
  Interventions: Drug: MK-5108
- MK-5108 1800 mg BID (Panel 1) (Experimental): Participants receive 1800 mg of MK-5108 orally BID the first 2 days of a 14-day cycle (cycle extended to 21 days if ≥Grade 2 toxicity observed).
  Interventions: Drug: MK-5108
- MK-5108 100 mg BID + 60 mg/m^2 Docetaxel (Panel 2) (Experimental): Participants receive 100 mg of MK-5108 orally BID in combination with 60 mg/m^2 Docetaxel administered intravenously (IV) the first 2 days of a 21-day cycle.
  Interventions: Drug: MK-5108; Drug: docetaxel
- MK-5108 150 mg BID + 60 mg/m^2 Docetaxel (Panel 2) (Experimental): Participants receive 150 mg of MK-5108 orally BID in combination with 60 mg/m^2 Docetaxel administered IV the first 2 days of a 21-day cycle.
  Interventions: Drug: MK-5108; Drug: docetaxel
- MK-5108 225 mg BID + 60 mg/m^2 Docetaxel (Panel 2) (Experimental): Participants receive 150 mg of MK-5108 orally BID in combination with 60 mg/m^2 Docetaxel administered IV the first 2 days of a 21-day cycle.
  Interventions: Drug: MK-5108; Drug: docetaxel
- MK-5108 100 mg BID + 60 mg/m^2 Docetaxel (Crossover) (Experimental): After receiving treatment in Panel 1, one participant crossed over to Panel 2 per protocol following disease progression to receive 100 mg of MK-5108 orally BID in combination with 60 mg/m^2 Docetaxel administered IV the first 2 days of a 21-day cycle.
  Interventions: Drug: MK-5108; Drug: docetaxel
- MK-5108 150 mg BID + 60 mg/m^2 Docetaxel (Crossover) (Experimental): After receiving treatment in Panel 1, participants crossed over to Panel 2 per protocol following disease progression to receive 150 mg of MK-5108 orally BID in combination with 60 mg/m^2 Docetaxel administered IV the first 2 days of a 21-day cycle.
  Interventions: Drug: MK-5108; Drug: docetaxel

INTERVENTIONS:
Drug: MK-5108 — MK-5108 will be administered orally, every 12 hours (Q12H) during the first 2 days of each cycle. Cycle length will be 14-21 days in Panel 1 and 21 days in Panel 2.
Drug: docetaxel — Docetaxel will be administered intravenously (I.V.) at a dose of 60 mg/m^2 Q12H during the first 2 days of each 21-day cycle.
  Other Names: Taxotere
  Arms: MK-5108 100 mg BID + 60 mg/m^2 Docetaxel (Crossover); MK-5108 100 mg BID + 60 mg/m^2 Docetaxel (Panel 2); MK-5108 150 mg BID + 60 mg/m^2 Docetaxel (Crossover); MK-5108 150 mg BID + 60 mg/m^2 Docetaxel (Panel 2); MK-5108 225 mg BID + 60 mg/m^2 Docetaxel (Panel 2)

SUMMARY:
This study will investigate the safety, side effects and how well the body tolerates MK-5108 as well as determine different doses of MK-5108 in participants with advanced and/or refractory solid tumors. The corresponding primary hypotheses of this study are that 1) administration of oral MK-5108 (twice daily for 2 out of 14-21 days) to participants with advanced and/or refractory solid tumors will be safe and tolerable, and that 2) the spectrum of side effects observed in these participants after administration of oral MK-5108 alone and in combination with docetaxel will be dose-dependent and allow for definition of a maximum tolerated dose (MTD).

ELIGIBILITY:
Inclusion Criteria:

- Participant has a histologically-confirmed metastatic or locally advanced solid tumor that has failed to respond to standard therapy or progressed with standard therapy

Exclusion Criteria:

* Participant has had chemotherapy, radiotherapy or biological therapy within 4 weeks prior to study start or has not recovered from adverse events caused by therapy more than 4 weeks earlier
* Participant is currently participating or has participated in a study with an investigational compound or device within 4 weeks prior to signing informed consent
* Participant has received more than 2 courses of chemotherapy for metastatic disease
* Participant has had prolonged neutropenia or neutropenia with fever from previous chemotherapy treatment
* Participant has a primary central nervous system tumor
* Participant is a regular or recreational user of any illicit drugs or has a recent history within the last year of drug or alcohol abuse
* Participant is pregnant, breastfeeding or planning to have children during the study
* Participant is Human Immunodeficiency Virus (HIV) positive
* Participant has a history of Hepatitis B or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-03-27 (Actual); Primary Completion 2011-04-04 (Actual); Study Completion 2011-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Amin M, Minton SE, LoRusso PM, Krishnamurthi SS, Pickett CA, Lunceford J, Hille D, Mauro D, Stein MN, Wang-Gillam A, Trull L, Lockhart AC. A phase I study of MK-5108, an oral aurora a kinase inhibitor, administered both as monotherapy and in combination with docetaxel, in patients with advanced or refractory solid tumors. Invest New Drugs. 2016 Feb;34(1):84-95. doi: 10.1007/s10637-015-0306-7. Epub 2015 Dec 1. PMID 26620496

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 35 participants were enrolled and treated in this study. 14 enrolled into Panel 1 and received MK-5108 monotherapy. An additional 4 enrolled into Panel 1 and received MK-5108 as monotherapy prior to crossing over to Panel 2 and receiving MK-5108 with docetaxel. 17 enrolled into Panel 2 and received only the combination of MK-5108 and docetaxel.
Groups:
- MK-5108 200 mg BID (Panel 1): Participants received 200 mg of MK-5108 orally twice daily (BID) the first 2 days of a 14-day cycle (cycle extended to 21 days if ≥Grade 2 toxicity observed).
- MK-5108 400 mg BID (Panel 1): Participants received 400 mg of MK-5108 orally BID the first 2 days of a 14-day cycle (cycle extended to 21 days if ≥Grade 2 toxicity observed).
- MK-5108 800 mg BID (Panel 1): Participants received 800 mg of MK-5108 orally BID the first 2 days of a 14-day cycle (cycle extended to 21 days if ≥Grade 2 toxicity observed).
- MK-5108 1200 mg BID (Panel 1): Participants received 1200 mg of MK-5108 orally BID the first 2 days of a 14-day cycle (cycle extended to 21 days if ≥Grade 2 toxicity observed).
- MK-5108 1500 mg BID (Panel 1): Participants received 1500 mg of MK-5108 orally BID the first 2 days of a 14-day cycle (cycle extended to 21 days if ≥Grade 2 toxicity observed).
- MK-5108 1800 mg BID (Panel 1): Participants received 1800 mg of MK-5108 orally BID the first 2 days of a 14-day cycle (cycle extended to 21 days if ≥Grade 2 toxicity observed).
Period: Panel 1 + Panel 2
Arm/Group | MK-5108 200 mg BID (Panel 1) | MK-5108 400 mg BID (Panel 1) | MK-5108 800 mg BID (Panel 1) | MK-5108 1200 mg BID (Panel 1) | MK-5108 1500 mg BID (Panel 1) | MK-5108 1800 mg BID (Panel 1) | MK-5108 100 mg BID + 60 mg/m^2 Docetaxel (Panel 2) | MK-5108 150 mg BID + 60 mg/m^2 Docetaxel (Panel 2) | MK-5108 225 mg BID + 60 mg/m^2 Docetaxel (Panel 2) | MK-5108 100 mg BID + 60 mg/m^2 Docetaxel (Crossover) | MK-5108 150 mg BID + 60 mg/m^2 Docetaxel (Crossover)
Started | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 5 | 0 | 0
Crossed Over to Panel 2 Due to PD | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 5 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Progressive Disease (PD) | 3 | 2 | 2 | 3 | 3 | 3 | 5 | 4 | 4 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Crossover Participants
Arm/Group | MK-5108 200 mg BID (Panel 1) | MK-5108 400 mg BID (Panel 1) | MK-5108 800 mg BID (Panel 1) | MK-5108 1200 mg BID (Panel 1) | MK-5108 1500 mg BID (Panel 1) | MK-5108 1800 mg BID (Panel 1) | MK-5108 100 mg BID + 60 mg/m^2 Docetaxel (Panel 2) | MK-5108 150 mg BID + 60 mg/m^2 Docetaxel (Panel 2) | MK-5108 225 mg BID + 60 mg/m^2 Docetaxel (Panel 2) | MK-5108 100 mg BID + 60 mg/m^2 Docetaxel (Crossover) | MK-5108 150 mg BID + 60 mg/m^2 Docetaxel (Crossover)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (Participant originally treated in MK-5108 400 mg BID (Panel 1) in Period 1) | 3 (3 participants originally treated with 1500 (2) and 1800 mg (1) MK-5108 in Panel 1 Period 1)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-5108 200 mg BID (Panel 1) | MK-5108 400 mg BID (Panel 1) | MK-5108 800 mg BID (Panel 1) | MK-5108 1200 mg BID (Panel 1) | MK-5108 1500 mg BID (Panel 1) | MK-5108 1800 mg BID (Panel 1) | MK-5108 100 mg BID + 60 mg/m^2 Docetaxel (Panel 2) | MK-5108 150 mg BID + 60 mg/m^2 Docetaxel (Panel 2) | MK-5108 225 mg BID + 60 mg/m^2 Docetaxel (Panel 2) | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 5 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (11.4) | 57.0 (7.8) | 75.3 (9.1) | 58.0 (15.7) | 54.3 (7.5) | 61.0 (2.0) | 58.0 (15.1) | 57.3 (15.7) | 59.8 (8.9) | 59.1 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 2 | 0 | 1 | 4 | 2 | 3 | 15
  Male | 1 | 3 | 2 | 1 | 3 | 2 | 2 | 4 | 2 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the Sponsor's product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition which is temporally associated with the use of the Sponsor's product, was also an AE. The number of participants who experienced an AE was reported for each dose level group.
Time Frame: From Day 1 of study treatment until 30 days following the last dose of study treatment (up to 577 days)
Population: All participants that received one or more doses of study medication. Four participants who received MK-5108 monotherapy in Panel 1 and then crossed over to receive combination treatment in Panel 2 (Crossover) were included in both respective treatment groups and AEs were reported according to treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-5108 200 mg BID (Panel 1) | MK-5108 400 mg BID (Panel 1) | MK-5108 800 mg BID (Panel 1) | MK-5108 1200 mg BID (Panel 1) | MK-5108 1500 mg BID (Panel 1) | MK-5108 1800 mg BID (Panel 1) | MK-5108 100 mg BID + 60 mg/m^2 Docetaxel (Panel 2) | MK-5108 150 mg BID + 60 mg/m^2 Docetaxel (Panel 2) | MK-5108 225 mg BID + 60 mg/m^2 Docetaxel (Panel 2) | MK-5108 100 mg BID + 60 mg/m^2 Docetaxel (Crossover) | MK-5108 150 mg BID + 60 mg/m^2 Docetaxel (Crossover)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 5 | 1 | 3
Participants | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 5 | 1 | 3

2. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLTs were AEs considered related to study drug that prevented escalation of the drug dose. Hematologic DLTs included any Grade 5 hematologic toxicity, Grade 4 neutropenia lasting for ≥7 days in duration, Grade 3 or Grade 4 neutropenia with fever >38.5°C and/or infection requiring antibiotic or anti-fungal treatment, and Grade 4 thrombocytopenia (≤25.0 x 10^9/L). Non-hematologic DLT was defined as any Grade 3, 4, or 5 non-hematologic toxicity, with the specific exceptions of: Grade 3 nausea or Grade 3 vomiting, Grade 3 diarrhea, or Grade 3 dehydration occurring in the setting of inadequate compliance with supportive care and lasting for <48 hours, alopecia, inadequately treated hypersensitivity reactions, or Grade 3 elevated transaminases of ≤1 week in duration. Any drug-related AE leading to a dose modification of MK-5108, or any unresolved drug-related toxicity persisting>6 weeks, was also considered a DLT.
Time Frame: Day 1 to Day 21 of study treatment (Cycle 1 for Panel 1, Panel 2, or Crossover)
Population: All participants that received one or more doses of study medication. Participants who received MK-5108 monotherapy in Panel 1 and then crossed over to receive combination treatment in Panel 2 (Crossover) were included in both respective treatment groups and DLTs were reported according to treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-5108 200 mg BID (Panel 1) | MK-5108 400 mg BID (Panel 1) | MK-5108 800 mg BID (Panel 1) | MK-5108 1200 mg BID (Panel 1) | MK-5108 1500 mg BID (Panel 1) | MK-5108 1800 mg BID (Panel 1) | MK-5108 100 mg BID + 60 mg/m^2 Docetaxel (Panel 2) | MK-5108 150 mg BID + 60 mg/m^2 Docetaxel (Panel 2) | MK-5108 225 mg BID + 60 mg/m^2 Docetaxel (Panel 2) | MK-5108 100 mg BID + 60 mg/m^2 Docetaxel (Crossover) | MK-5108 150 mg BID + 60 mg/m^2 Docetaxel (Crossover)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 5 | 1 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: From Day 1 of study treatment until 30 days following the last dose of study treatment (up to 577 days)
Description: All participants that received one or more doses of study medication. Four participants who received MK-5108 monotherapy in Panel 1 and then crossed over to receive combination treatment in Panel 2 (Crossover) were included in both respective treatment groups and AEs were reported according to treatment received.
Groups:
- MK-5108 100 mg BID + 60 mg/m2 Docetaxel (Panel 2): Participants received 100 mg of MK-5108 orally BID in combination with 60 mg/m^2 Docetaxel administered intravenously (IV) the first 2 days of a 21-day cycle.
- MK-5108 150 mg BID + 60 mg/m2 Docetaxel (Panel 2): Participants received 150 mg of MK-5108 orally BID in combination with 60 mg/m^2 Docetaxel administered IV the first 2 days of a 21-day cycle.
- MK-5108 225 mg BID + 60 mg/m2 Docetaxel (Panel 2): Participants received 225 mg of MK-5108 orally BID in combination with 60 mg/m^2 Docetaxel administered IV the first 2 days of a 21-day cycle.
- MK-5108 100 mg BID + 60 mg/m2 Docetaxel (Crossover): After receiving treatment in Panel 1, one participant crossed over to Panel 2 per protocol following disease progression to receive 100 mg of MK-5108 orally BID in combination with 60 mg/m^2 Docetaxel administered IV the first 2 days of a 21-day cycle.
- MK-5108 150 mg BID + 60 mg/m2 Docetaxel (Crossover): After receiving treatment in Panel 1, participants crossed over to Panel 2 per protocol following disease progression to receive 150 mg of MK-5108 orally BID in combination with 60 mg/m^2 Docetaxel administered IV the first 2 days of a 21-day cycle.
Arm/Group | MK-5108 200 mg BID (Panel 1) | MK-5108 400 mg BID (Panel 1) | MK-5108 800 mg BID (Panel 1) | MK-5108 1200 mg BID (Panel 1) | MK-5108 1500 mg BID (Panel 1) | MK-5108 1800 mg BID (Panel 1) | MK-5108 100 mg BID + 60 mg/m2 Docetaxel (Panel 2) | MK-5108 150 mg BID + 60 mg/m2 Docetaxel (Panel 2) | MK-5108 225 mg BID + 60 mg/m2 Docetaxel (Panel 2) | MK-5108 100 mg BID + 60 mg/m2 Docetaxel (Crossover) | MK-5108 150 mg BID + 60 mg/m2 Docetaxel (Crossover)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 1/3 | 0/3 | 0/6 | 0/6 | 0/5 | 0/1 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 1/3 | 0/3 | 1/3 | 0/3 | 1/6 | 4/6 | 4/5 | 0/1 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 2/3 | 3/3 | 3/3 | 3/3 | 2/3 | 5/6 | 6/6 | 4/5 | 1/1 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-5108 200 mg BID (Panel 1) (N=3) | MK-5108 400 mg BID (Panel 1) (N=3) | MK-5108 800 mg BID (Panel 1) (N=3) | MK-5108 1200 mg BID (Panel 1) (N=3) | MK-5108 1500 mg BID (Panel 1) (N=3) | MK-5108 1800 mg BID (Panel 1) (N=3) | MK-5108 100 mg BID + 60 mg/m2 Docetaxel (Panel 2) (N=6) | MK-5108 150 mg BID + 60 mg/m2 Docetaxel (Panel 2) (N=6) | MK-5108 225 mg BID + 60 mg/m2 Docetaxel (Panel 2) (N=5) | MK-5108 100 mg BID + 60 mg/m2 Docetaxel (Crossover) (N=1) | MK-5108 150 mg BID + 60 mg/m2 Docetaxel (Crossover) (N=3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-5108 200 mg BID (Panel 1) (N=3) | MK-5108 400 mg BID (Panel 1) (N=3) | MK-5108 800 mg BID (Panel 1) (N=3) | MK-5108 1200 mg BID (Panel 1) (N=3) | MK-5108 1500 mg BID (Panel 1) (N=3) | MK-5108 1800 mg BID (Panel 1) (N=3) | MK-5108 100 mg BID + 60 mg/m2 Docetaxel (Panel 2) (N=6) | MK-5108 150 mg BID + 60 mg/m2 Docetaxel (Panel 2) (N=6) | MK-5108 225 mg BID + 60 mg/m2 Docetaxel (Panel 2) (N=5) | MK-5108 100 mg BID + 60 mg/m2 Docetaxel (Crossover) (N=1) | MK-5108 150 mg BID + 60 mg/m2 Docetaxel (Crossover) (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 2 (6) | 5 (9) | 2 (8) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 1 (1) | 4 (17) | 2 (3) | 3 (8) | 0 (0) | 1 (3)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 3 (23) | 1 (4) | 1 (2) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (12) | 5 (10) | 3 (7) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal wall cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 3 (3) | 2 (2) | 4 (7) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 2 (6) | 2 (5) | 1 (1) | 1 (3)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 2 (2) | 1 (1) | 2 (8) | 2 (2) | 1 (1) | 4 (7) | 3 (3) | 3 (3) | 1 (2) | 2 (2)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 4 (8) | 2 (3) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (5) | 2 (4) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 3 (7)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0) | 1 (3) | 3 (4) | 2 (3) | 0 (0) | 4 (12) | 4 (7) | 3 (5) | 0 (0) | 3 (5)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Local swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Puncture site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucocutaneous candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incision site complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Bilirubin conjugated increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood bicarbonate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 1 (2) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glucose urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostatic specific antigen increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (3) | 1 (2) | 1 (1) | 1 (1) | 3 (3) | 2 (3) | 3 (5) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 1 (2) | 2 (3) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3) | 2 (4) | 1 (3) | 1 (2) | 4 (11) | 3 (17) | 2 (8) | 0 (0) | 2 (10)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (7) | 0 (0) | 0 (0) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 2 (6) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (6)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (2) | 1 (3) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nodule on extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 2 (3) | 1 (2) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (4)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (6) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (8) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parosmia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Emotional distress (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mood swings (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Penile oedema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (4) | 2 (3) | 0 (0) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (9) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lichenification (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines.